CLINICAL TRIAL: NCT00002922
Title: Phase II Evaluation of Paclitaxel Infusion in Advanced (Recurrent or Metastatic) Squamous Cell Carcinoma of the Head and Neck
Brief Title: Paclitaxel in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065327; E-3395
Record Dates: First submitted 1999-11-01; First posted 2004-07-07 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the response rate and toxic effects of paclitaxel by 96 hour continuous infusion in chemotherapy naive and chemotherapy exposed patients with recurrent or metastatic squamous cell carcinoma of the head and neck.

OUTLINE: Patients receive paclitaxel as a 96 hour continuous IV infusion. Courses repeat every 3 weeks for a maximum of 12 courses. Patients with disease progression after 2 courses or with unacceptable toxicity at any time are removed from study.

PROJECTED ACCRUAL: Approximately 109 patients will be accrued for this study over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the head and neck (including nasopharynx) that is considered incurable with surgery or radiation therapy Bidimensionally measurable disease Patients whose only site of measurable disease is within a previous radiation port must have documented progressive disease or biopsy-proven recurrence after the completion of radiotherapy No uncontrolled CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Calcium normal No history of hypercalcemia Cardiovascular: No history of ventricular arrhythmias or symptomatic bradyarrhythmia Other: No significant detectable infection Not pregnant or nursing No other active malignancies Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior interleukin-2, interferons, and monoclonal antibodies allowed Recovered from prior therapy Chemotherapy: Prior paclitaxel infusion no greater than 24 hours for recurrent or metastatic disease required Endocrine therapy: Not specified Radiotherapy: Recovered from prior radiotherapy Surgery: Recovered from any prior major surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-02-21 (Actual); Primary Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (24):
- United States (23):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - New England Medical Center Hospital, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Langer CJ, Li Y, Jennings T, DeConti RC, Nair S, Cohen RB, Forastiere AA; Eastern Cooperative Oncology Group. Phase II evaluation of 96-hour paclitaxel infusion in advanced (recurrent or metastatic) squamous cell carcinoma of the head and neck (E3395): a trial of the Eastern Cooperative Oncology Group. Cancer Invest. 2004;22(6):823-31. doi: 10.1081/cnv-200039628. PMID 15641479